CLINICAL TRIAL: NCT05745558
Title: PREoPerAtive pREhabilitation in Patients With Head and Neck Cancer or Liver Cancer (PREPARE)
Acronym: PREPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Rijndam Revalidatiecentrum (Unknown); Capri Hartrevalidatie (Unknown)
Responsible Party: Principal Investigator, Roeland F. de Wilde, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL 80823.078.22
Record Dates: First submitted 2023-02-06; First posted 2023-02-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cancer Liver; Cancer Head Neck
MeSH Terms: conditions — Carcinoma, Hepatocellular; Head and Neck Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Prospective Cohort Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): A 3-to-6-week prehabilitation program consisting of training and nutritional, smoking cessation and psychosocial counselling.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — The prehabilitation program consists of 4 components:
  1. Fitness training led by a physiotherapist. The patients will receive personalized training schedules to perform at home. The training sessions focus on improving aerobic fitness (biking or walking) and muscle strength (specific exercises for the different patient groups) and respiratory exercises aimed to relax.
  2. Nutritional counseling led by a dietician. All patients will be offered an intake with a dietician (60 min) to discuss current eating habits and give personalized advices. Based on indication, patients will receive follow-up consults.
  3. Smoking cessation counseling led by a trained social worker. For patients that are currently smoking, a social worker will offer counseling sessions to coach the patient in the process of smoking cessation.
  4. Psychosocial counseling led by a psychologist. All patients will be offered counselling by a psychologist.

SUMMARY:
The objective of this study is to determine the feasibility (main aim) and effectiveness (secondary aim) of a prehabilitation program in patients with head and neck cancer or liver cancer. Participating patients will participate in a 3-to-6 week rehabilitation program consisting of training and nutritional, smoking cessation and psychosocial counselling.

DETAILED DESCRIPTION:
In patients diagnosed with head and neck cancer (HNC) or liver cancer, (major) surgery is the standard of care. Nevertheless, surgery may result in complications that have a substantial impact on the physical and psychological state of the patient. Detrimental postoperative outcomes are influenced by unhealthy lifestyle behaviors such as a sedentary lifestyle, smoking and malnutrition. Prehabilitation programs focusing on these lifestyle aspects have been suggested as a promising intervention to improve pre- and postoperative outcomes. Therefore, the obective of this study is to determine the feasibility (main aim) and effectiveness (secondary aim) of a prehabilitation program in patients with HNC or liver cancer

This study concerns a prospective cohort study in 60 patients with HNC or liver cancer that participate in a 3 to 6-week pilot prehabilitation program consisting of training and nutritional, smoking cessation and psychosocial counselling.

Data on feasibility (program satisfaction, program compliance and percentage of patients willing to participate in the prehabilitation program) and effectiveness (e.g. complications, health status, compliance to healthy lifestyle) is collected at three time points (pre- and post the prehabilitation program and 30 days post-surgery).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of head and neck cancer or liver cancer
* Scheduled for surgery in Erasmus MC
* Provision of written informed consent
* Only patient with a waiting time of at least 3 weeks till surgery can participate in this study

Exclusion Criteria:

* Patients that do not understand the Dutch language
* Patients with severe physical or psychological comorbidities that limit participation in the prehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Program satisfaction | At completion of the prehabilitation program (3-6 weeks after baseline)
  Self-designed questionnaire score (score between 1-10, higher score means higher satisfaction)
Program compliance | At completion of the prehabilitation program (3-6 weeks after baseline)
  Number of sessions that patient participates in the fitness training, the counselling on nutrition, smoking cessation and psychosocial sessions will be registered.
Percentage of patients willing to participate in prehabilitation program | At completion of the prehabilitation program (3-6 weeks after baseline)
  It will be registered which patient are willing and not willing to participate

SECONDARY OUTCOMES:
Frailty | Outcomes will be collected twice: at baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Groningen Frailty Score questionnaire score: score of 0-15, a GFI score of four or greater is considered the cut-off point for frailty
Functional capacity | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  6-minute walk test: meters walked in 6 minutes time
Physical activity level | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  ActiGraph GTx3+ accelerometer: average time per day (min) spend in moderate-to-vigorous activity, light physical activity and sedentary behaviour
Hand grip strength | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Hand dynamometer (kg)
Quadriceps strength | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Biodex dynamometer (Peak torque to body weight extension + Work fatigue)
Nutritional status | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Short Nutritional Assessment Questionnaire (SNAQ) score (range 4-20, lower score means higher risk of malnutrition)
Body composition | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Weight scale (kg)
Health status | At baseline, at completion of the prehabilitation program (3-6 weeks after baseline), 30 days post surgery
  EuroQol-5D (EQ5D) questionnaire score (0-1, the maximum score of 1 indicates the best health state)
Anxiety and Depression | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Hospital Anxiety and Depression Scale questionnaire score (0-21, higher scores denotes risk of anxiety or depression
Self-efficacy | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  General Self Efficacy Scale questionnaire score (10-40, with a higher score indicating more self-efficacy
Self-reported smoking behaviour | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Self-designed questionnaire (smoking yes/no)
Smoking behaviour | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  carbon monoxide breath analyser (CO ppm + % COhb)
Alcohol consumptiom | At baseline and at completion of the prehabilitation program (3-6 weeks after baseline)
  Five shot questionnaire score (0-7, a higher score indicates possible alcohol misuse)
Length of hospital stay | 30 days post surgery
  Registrered in patient file (length in days)
Complications Clavien Dindo grade ≥3 in first 30 days | 30 days post surgery
  Registrered in patient file (number of complications and clavien dindo grade)
Readmission rate in first 30 days | 30 days post surgery
  Number and reason for readmissions in first 30 days
Age | Baseline
  Age in years
Sex | Baseline
  Female/male/other
Medical diagnosis | Baseline
  Medical diagnosis for surgery
Educational level | Baseline
  Single-item question (high, middle, low educated)
Marital status | Baseline
  Single-item question (Partnered/ unpartnered)
Work status | Baseline
  Single-item question (employed/unemployed)

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No